CLINICAL TRIAL: NCT02224053
Title: A Phase I, Fixed Sequence, Open-label, Study to Assess the Pharmacokinetics of AZD9291 in Healthy Male Volunteers When a Single Oral Dose of AZD9291 80 mg is Administered Alone and in Combination With Omeprazole
Brief Title: Drug-Drug Interaction Study With AZD9291 and Omeprazole in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D5160C00010
Record Dates: First submitted 2014-08-20; First posted 2014-08-25 (Estimated); Results first posted 2015-12-31 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Healthy Volunteer
Keywords: oncology, cancer, non small cell lung cancer, anticancer druge, omeprazole, healthy volunteer
MeSH Terms: conditions — Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- AZD9291 and omeprazole (Experimental): Sequential treatments of AZD9291 + omeprazole followed by AZD9291 alone, with a washout period in between.
  Interventions: Procedure: Pharmacokinetic sampling - AZD9291; Drug: AZD9291 tablet dosing; Drug: Omeprazole tablet dosing; Procedure: Pharmacokinetic sampling - AZ5140 and AZ7550

INTERVENTIONS:
Procedure: Pharmacokinetic sampling - AZD9291 — Blood sampling to measure AZD9291
Drug: AZD9291 tablet dosing — AZD9291 80mg tablet taken on Day 5 in Period 1 and Day 1 in Period 2.
Drug: Omeprazole tablet dosing — Omeprzole taken from Days 1 to 5 in Period 1.
Procedure: Pharmacokinetic sampling - AZ5140 and AZ7550 — Blood samples to measure levels of AZ5140 and AZ7550

SUMMARY:
This is a Phase 1, open-label, 2-period fixed sequence design to evaluate the interaction of AZD9291 with omeprazole in approximately 50 healthy, adult male volunteers. Volunteers will receive Treatment A (AZD9291 and omeprazole) in Period 1 and Treatment B (AZD9291 only) in Period 2. The dose of AZD9291 in Period 1 and the dose of AZD9291 in Period 2 will be separated by a washout of at least 21 days (the washout will not be more than 5 weeks). The study will be performed at up to 2 sites in the USA and will assess the effect of omeprazole (proton pump inhibitor) on AZD9291 exposure

ELIGIBILITY:
For inclusion in the study volunteers must fulfil the following criteria.

1. Provision of signed and dated informed consent prior to any study-specific procedures.
2. Healthy male volunteers aged 18 to 55 years. (Healthy as determined by medical history, physical examination, laboratory parameters, ECG, and eye examination performed before the first administration of investigational product.)
3. Body mass index between 19 and 30 kg/m2, and body weight between 50 kg and 100 kg, inclusive.
4. Veins suitable for cannulation or repeated venepuncture.
5. Volunteers must be willing to use reliable methods of contraception (condom and spermicide), even if their partners are postmenopausal, surgically sterile, or using an effective hormonal method of contraception or intrauterine coil. In addition, volunteers must agree to continue to take similar contraceptive precautions and avoid sperm donation for 6 months after the last administration of AZD9291.

Volunteers must not enter the study if any of the following exclusion criteria are fulfilled:

1. Involvement in the planning and/or conduct of the study (applies to both AstraZeneca and Quintiles staff).
2. Previous enrollment in the present study.
3. History of any clinically significant disease or disorder which, in the opinion of the Investigator, may either put the healthy volunteer at risk because of participation in the study, or influence the results or the healthy volunteer's ability to participate in the study.
4. History or presence of gastrointestinal, hepatic, or renal disease or surgical procedure or any other condition known to interfere with the absorption, distribution, metabolism, or excretion of drugs.
5. Any clinically significant abnormalities in physical examination, vital signs (supine blood pressure >140 mmHg systolic, >90 mmHg diastolic, or pulse rate ≤35 or ≥100 beats per minute), or clinical laboratory assessment as judged by the Investigator.
6. Acute illness, surgical procedures, or trauma from within 2 weeks before enrollment until first administration of investigational product (IP).
7. Volunteers who have received live or live-attenuated vaccine in the 2 weeks prior to dosing.
8. Volunteers with active malignancy or neoplastic disease in the previous 12 months.
9. A suspected/manifested infection according to International Airline Transportation Association (IATA) Categories A and B infectious substances.
10. Positive results on screening tests for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody, or human immunodeficiency virus (HIV).
11. Any clinically important abnormalities in rhythm, conduction, or morphology of resting ECG, as judged by the Investigator.
12. Known or suspected history of significant drug abuse as judged by the Investigator.
13. Positive screen for drugs of abuse or cotinine (nicotine level above 400 ng/mL) at screening or positive screen for alcohol, drugs of abuse, or cotinine on admission in Period 1 or Period 2.
14. History of alcohol abuse or excessive intake of alcohol, defined as regular weekly intake of greater than 21 units of alcohol in men (Note: 1 unit=25 mL spirits, 125 mL wine, or 250 mL beer or lager).
15. History of severe allergy/hypersensitivity or ongoing allergy/hypersensitivity, as judged by the Investigator, or history of hypersensitivity to AZD9291, its excipients, or drugs with a similar chemical structure or class.
16. History of hypersensitivity to omeprazole, its excipients, or drugs with a similar chemical structure or class.
17. Use of any prescribed or nonprescribed medication, including drugs with hepatic enzyme-altering properties, such as St John's Wort, antacids, analgesics, herbal remedies, vitamins, and minerals during the 4 weeks (or longer depending on the medication's half-life) prior to the first administration of AZD9291 is not permitted. Occasional use of paracetamol (acetaminophen) and nonsteroidal nasal decongestant is permitted at the discretion of the Investigator.
18. Any intake of grapefruit, grapefruit juice, Seville oranges, Seville orange marmalade, or other products containing grapefruit or Seville oranges within 7 days of the first administration of IP.
19. Blood donation within 1 month of screening or any blood donation/blood loss greater than 500 mL during the 3 months prior to screening.
20. Use of another new chemical entity (defined as a compound which has not been approved for marketing) or participation in any other clinical study (including methodology studies where no drugs were given) within 3 months of the first administration of IP in this study.
21. Current smokers or those who have smoked or used nicotine products within the previous 3 months.
22. Planned inpatient surgery, dental procedure, or hospitalisation during the study.

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 136 (Actual)
Dates: Start 2014-09; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Serban Ghiorghiu, MSD, Study Director — AstraZeneca
Locations (2):
- United States (2):
  - Research Site, Overland Park, Kansas
  - Research Site, Minneapolis, Minnesota

REFERENCES:
- [Derived] Vishwanathan K, Dickinson PA, Bui K, Cassier PA, Greystoke A, Lisbon E, Moreno V, So K, Thomas K, Weilert D, Yap TA, Plummer R. The Effect of Food or Omeprazole on the Pharmacokinetics of Osimertinib in Patients With Non-Small-Cell Lung Cancer and in Healthy Volunteers. J Clin Pharmacol. 2018 Apr;58(4):474-484. doi: 10.1002/jcph.1035. Epub 2017 Nov 26. PMID 29178442

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled: 3 September 2014 Last Subject Last Visit: 5 January 2015 Study was performed at 2 sites in the USA.
Pre-assignment Details: 136 subjects were enrolled (signed informed consent). Subjects were assigned to treatment if they met all the inclusion and none of the exclusion criteria.
  68 subjects were enolled but failed inclusion/exclusion criteria and so were not eligible to be assigned treatment.
  The remaining 68 subjects started period 1 and received treatment.
Groups:
- AZD9291 and Omeprazole: Sequential treatments periods of AZD9291 + omeprazole (including a washout) followed by AZD9291 alone.
Period: AZD9291 and Omeprazole Co-administration
Arm/Group | AZD9291 and Omeprazole
Started | 68
Completed | 47
Not Completed | 21
Not completed — Exceeding PK limits after Period 1 | 11
Not completed — Protocol Violation | 4
Not completed — Adverse Event | 3
Not completed — Withdrawal by Subject | 1
Not completed — Protocol non-compliance | 2
Period: AZD9291 Alone
Arm/Group | AZD9291 and Omeprazole
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | AZD9291 and Omeprazole
Number analyzed (Participants) | 68
Age, Continuous [Mean (Standard Deviation); unit: Years] | 34.0 (11.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 68

OUTCOME MEASURES:

1. Primary Outcome: AUC of AZD9291
Description: Area under the plasma concentration-time curve from zero to infinity for AZD9291
Time Frame: PK samples collected in both period 1 and 2 at pre-dose, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72, 120, 168, 216, 336, and 504 hours post AZD9291 dose
Population: Pharmacokinetic population - all subjects who received at least 1 dose of AZD9291 and had at least 1 postdose PK measurement without important protocol deviations/violations or events thought to significantly affect the PK of the investigational product
Measure: Geometric Mean (Full Range); unit: nM.h
Groups:
- AZD9291 and Omeprazole Co-administration: Once daily dosing of omeprazole 40 mg on Days 1 to 5 and AZD9291 80 mg single oral dose on Day 5 (Period 1).
- AZD9291 Alone: AZD9291 80 mg single oral dose on Day 1 (Period 2)
Arm/Group | AZD9291 and Omeprazole Co-administration | AZD9291 Alone
Number analyzed (Participants) | 53 | 47
nM.h | 6690 (28.8) [2340 to 10200] | 6269 (37.0) [2670 to 14200]
Statistical Analysis 1: Comparison: AZD9291 and Omeprazole Co-administration vs AZD9291 Alone; Study sized so experiment-wise power for the 90% CIs of geometric mean ratios for both AUC and Cmax of AZD9291 being within 80% to 125% was 90% (95% for each parameter). Within subject CV assumed to be 23%. 5% change in exposure also assumed; Test type: Non-Inferiority or Equivalence — 90% CIs of geometric mean ratios being within 80% to 125%; Geometric mean ratio = 106.66, 90% CI 2-sided [100.26 to 113.46] — AZD9291+omeprazole / AZD9291 alone

2. Primary Outcome: Cmax of AZD9291
Description: Rate and extent of absorption of AZD9291 following single oral doses of AZD9291 tablet formulation by assessment of maximum plasma concentration (Cmax).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: nM
Arm/Group | AZD9291 and Omeprazole Co-administration | AZD9291 Alone
Number analyzed (Participants) | 57 | 47
nM | 127.8 (26.9) [47.6 to 200] | 126.1 (31.0) [49.0 to 200]
Statistical Analysis 1: Comparison: AZD9291 and Omeprazole Co-administration vs AZD9291 Alone; [analysis description as in outcome 1, analysis 1]; Test type: Non-Inferiority or Equivalence — 90% CIs of geometric mean ratios being within 80% to 125%; Geometric mean ratio = 101.65, 90% CI 2-sided [94.65 to 109.16] — AZD9291+omeprazole / AZD9291 alone

3. Secondary Outcome: AUC(0-t)
Description: Assessment of the PK of AZD9291 (parent compound), AZ5104 (metabolite) and AZ7550 (metabolite) using area under the plasma concentration curve from zero extrapolated to o the time of the last quantifiable concentration, AUC(0-t)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: nM.h
Arm/Group | AZD9291 and Omeprazole Co-administration | AZD9291 Alone
Number analyzed (Participants) | 53 | 47
nM.h
  AZD9291 | 6673 [2340 to 10200] | 6249 [2660 to 14100]
  AZ5104 | 546.5 [226 to 939] | 539.2 [230 to 1110]
  AZ7550 | 520.0 [208 to 1010] | 560.0 [300 to 942]

4. Secondary Outcome: AUC(0-72)
Description: Assessment of the PK of AZD9291 (parent compound), AZ5104 (metabolite) and AZ7550 (metabolite) using area under the plasma concentration curve from time zero to 72 hours, AUC(0-72)
Time Frame: PK samples collected in both period 1 and 2 at pre-dose, 1, 2, 3, 4, 5, 6, 7, 8, 10, 12, 24, 48, 72 hours post AZD9291 dose.
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: nM.h
Arm/Group | AZD9291 and Omeprazole Co-administration | AZD9291 Alone
Number analyzed (Participants) | 54 | 47
nM.h
  AZD9291 | 4404 [1710 to 6410] | 4106 [1760 to 7530]
  AZ5104 | 301.5 [151 to 589] | 304.0 [153 to 540]
  AZ7550 | 216.5 [82.1 to 398] | 231.3 [100 to 445]

5. Secondary Outcome: Tmax
Description: Assessment of the PK of AZD9291 (parent compound), AZ5104 (metabolite) and AZ7550 (metabolite) using time to reach maximum plasma concentration, tmax
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | AZD9291 and Omeprazole Co-administration | AZD9291 Alone
Number analyzed (Participants) | 57 | 47
h
  AZD9291 | 6 [5 to 48.08] | 6 [3 to 12.1]
  AZ5104 | 8 [5 to 72.12] | 7 [4 to 48.05]
  AZ7550 | 10 [5 to 72.42] | 10 [5 to 71.77]

6. Secondary Outcome: Tlag
Description: Assessment of the PK of AZD9291 (parent compound), AZ5104 (metabolite) and AZ7550 (metabolite) using lag time before observation of quantifiable analyte concentrations in plasma, tlag
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: h
Arm/Group | AZD9291 and Omeprazole Co-administration | AZD9291 Alone
Number analyzed (Participants) | 57 | 47
h
  AZD9291 | 0.00 [0.00 to 0.00] | 0.00 [0.00 to 0.00]
  AZ5104 | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 1.00]
  AZ7550 | 0.00 [0.00 to 2.00] | 0.00 [0.00 to 1.00]

7. Secondary Outcome: t(1/2)
Description: Assessment of the PK of AZD9291 (parent compound), AZ5104 (metabolite) and AZ7550 (metabolite) using the terminal half-life, t(1/2)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: h
Arm/Group | AZD9291 and Omeprazole Co-administration | AZD9291 Alone
Number analyzed (Participants) | 53 | 47
h
  AZD9291 | 58.99 [39.2 to 77.1] | 63.60 [52.3 to 80.4]
  AZ5104 | 51.06 [31.1 to 85.4] | 54.47 [34.5 to 87.7]
  AZ7550 | 71.34 [47.0 to 106] | 72.16 [48.5 to 102]

8. Secondary Outcome: λz
Description: Assessment of the PK of AZD9291 (parent compound), AZ5104 (metabolite) and AZ7550 (metabolite) using the terminal rate constant, λz
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: 1/h
Arm/Group | AZD9291 and Omeprazole Co-administration | AZD9291 Alone
Number analyzed (Participants) | 53 | 47
1/h
  AZD9291 | 0.011748 [0.00899 to 0.0177] | 0.010898 [0.00862 to 0.0132]
  AZ5104 | 0.013577 [0.00812 to 0.0223] | 0.012722 [0.00790 to 0.0201]
  AZ7550 | 0.009718 [0.00656 to 0.0147] | 0.009606 [0.00677 to 0.0143]

9. Secondary Outcome: CL/F of AZD9291
Description: Assessment of the PK of AZD9291 using the apparent plasma clearance, CL/F
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: L/h
Arm/Group | AZD9291 and Omeprazole Co-administration | AZD9291 Alone
Number analyzed (Participants) | 53 | 47
L/h | 23.93 [15.6 to 68.4] | 25.55 [11.3 to 60.1]

10. Secondary Outcome: Vz/F of AZD9291
Description: Assessment of the PK of AZD9291 using the apparent volume of distribution, Vz/F
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: L
Arm/Group | AZD9291 and Omeprazole Co-administration | AZD9291 Alone
Number analyzed (Participants) | 53 | 47
L | 2037 [1280 to 3870] | 2343 [1250 to 5120]

11. Secondary Outcome: Cmax of AZ5104 and AZ7550
Description: Assessment of the PK of AZ5104 and AZ7550 (metabolites to AZD9291) using the maximum plasma concentration, Cmax
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: nM
Arm/Group | AZD9291 and Omeprazole Co-administration | AZD9291 Alone
Number analyzed (Participants) | 57 | 47
nM
  AZ5104 | 5.543 (26.9) [2.73 to 12.0] | 5.889 (31.0) [2.67 to 12.9]
  AZ7550 | 3.913 [1.68 to 7.98] | 4.402 [2.04 to 9.69]
Statistical Analysis 1: Comparison: AZD9291 and Omeprazole Co-administration vs AZD9291 Alone; AZ5104; Test type: Non-Inferiority or Equivalence — 90% CIs of geometric mean ratios being within 80% to 125%; Geometric mean ratio = 94.79, 90% CI 2-sided [88.77 to 101.21]
Statistical Analysis 2: Comparison: AZD9291 and Omeprazole Co-administration vs AZD9291 Alone; AZ7550; Test type: Non-Inferiority or Equivalence — 90% CIs of geometric mean ratios being within 80% to 125%; Geomteric mean ratio = 89.70, 90% CI 2-sided [83.89 to 95.91]

12. Secondary Outcome: AUC of AZ5104 and AZ7550
Description: Area under the plasma concentration-time curve from zero to infinity of AZ5104 and AZ7550 (metabolites to AZD9291)
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: nM.h
Arm/Group | AZD9291 and Omeprazole Co-administration | AZD9291 Alone
Number analyzed (Participants) | 53 | 47
nM.h
  AZ5104 | 556.6 (28.8) [231 to 948] | 550.7 (37.0) [245 to 1130]
  AZ7750 | 536.5 [231 to 1020] | 574.9 [309 to 955]
Statistical Analysis 1: Comparison: AZD9291 and Omeprazole Co-administration vs AZD9291 Alone; AZ5104; Test type: Non-Inferiority or Equivalence — 90% CIs of geometric mean ratios being within 80% to 125%; Geometric mean ratio = 102.32, 90% CI 2-sided [96.87 to 108.07] — AZD9291+omeprazole / AZD9291 alone
Statistical Analysis 2: Comparison: AZD9291 and Omeprazole Co-administration vs AZD9291 Alone; AZ7550; Test type: Non-Inferiority or Equivalence — 90% CIs of geometric mean ratios being within 80% to 125%; Geometric mean ratio = 94.03, 90% CI 2-sided [89.92 to 98.33]

13. Secondary Outcome: Parent to Metabolite Ratios of AZ5104 and AZ7550 Cmax
Description: Assessment of the PK of AZ5104 and AZ7550 Cmax using the parent (AZD9291) to metabolite ratios
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: Ratio
Arm/Group | AZD9291 and Omeprazole Co-administration | AZD9291 Alone
Number analyzed (Participants) | 57 | 47
Ratio
  AZ5104 | 0.04335 [0.0255 to 0.0873] | 0.04671 [0.0293 to 0.0908]
  AZ7550 | 0.03061 [0.0169 to 0.0530] | 0.03491 [0.0169 to 0.0708]

14. Secondary Outcome: Parent to Metabolite Ratios of AZ5104 and AZ7550 AUC
Description: Assessment of the PK of AZ5104 and AZ7550 AUC using the parent (AZD9291) to metabolite ratios
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Geometric Mean (Full Range); unit: Ratio
Arm/Group | AZD9291 and Omeprazole Co-administration | AZD9291 Alone
Number analyzed (Participants) | 53 | 47
Ratio
  AZ5104 | 0.08318 [0.0464 to 0.137] | 0.08785 [0.0587 to 0.133]
  AZ7550 | 0.08019 [0.0334 to 0.152] | 0.09166 [0.0424 to 0.207]

ADVERSE EVENTS:
Time Frame: AEs collected from the day prior to first dose of treatment (omeprazole) until the follow up visit, approximately 3 months.
Arm/Group | AZD9291 and Omeprazole Co-administration | AZD9291 Alone
Serious Adverse Events (participants affected / at risk) | 3/68 | 0/47
Other Adverse Events (participants affected / at risk) | 8/68 | 2/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9291 and Omeprazole Co-administration (N=68) | AZD9291 Alone (N=47)
Cholelithiasis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 1 (1) | 0 (0)
Transaminases increased (Investigations) | 2 (2) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 4% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AZD9291 and Omeprazole Co-administration (N=68) | AZD9291 Alone (N=47)
Headache (Nervous system disorders) | 5 (5) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 3 (3) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator (PI) agrees to collaborate on the contents and formation of any publication and to pay due consideration to comments and opinions offered. AstraZeneca have 30 days for final manuscript review and may require that submission for publication be delayed in order to file patent application.